CLINICAL TRIAL: NCT04205565
Title: A Randomized, Double-blind, Positive Drug/Placebo Parallel Controlled, Multicenter, Phase III Clinical Trial of L-oxiracetam Injection to Improve Memory and Cognitive Impairment in Patients With Craniocerebral Injury
Brief Title: Study on Clinical Effectiveness of L-Oxiracetam Injection
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing Yoko Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NJYK-L-ORCT-III
Record Dates: First submitted 2019-12-18; First posted 2019-12-19 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Craniocerebral Injury
Keywords: L-oxiracetam; Cognitive Impairment; Craniocerebral Injury
MeSH Terms: conditions — Craniocerebral Trauma; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- L-oxiracetam (Active Comparator)
  Interventions: Drug: Test group: L-oxiracetam Injection
- Oxiracetam (Active Comparator)
  Interventions: Drug: Control group: Oxiracetam Injection
- Plaecbo (Placebo Comparator)
  Interventions: Drug: Placebo group: Placebo Injection

INTERVENTIONS:
Drug: Test group: L-oxiracetam Injection — L-oxiracetam injection, 4 vials, once a day, IV. Placebo injection of oxiracetam, 6 vials, once a day, IV.
  Arms: L-oxiracetam
Drug: Control group: Oxiracetam Injection — Placebo injection of l-oxiracetam, 4 vials, once a day, IV. Oxiracetam injection, 6 vials, once a day, IV.
  Arms: Oxiracetam
Drug: Placebo group: Placebo Injection — Placebo injection of l-oxiracetam, 4 vials, once a day, IV. Placebo injection of oxiracetam, 6 vials, once a day, IV.
  Arms: Plaecbo

SUMMARY:
A randomized, double-blind, positive drug/placebo parallel controlled, multicenter, phase III clinical trial of L-oxiracetam injection to improve memory and cognitive Impairment in patients with craniocerebral injury.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old (including upper and lower limits), male or female
2. Craniocerebral injury meets all of the following conditions: This diagnosis has a clear head trauma, closed head injury, or head injury with cerebrospinal fluid ear leak and / or nasal leak and / or intracranial gas accumulation; MRI or CT confirmed intracranial hemorrhage above the cerebellum (including cerebral contusion, subarachnoid hemorrhage, epidural hematoma, subdural hemorrhage, intracranial hematoma, etc.), with or without transient coma; Craniocerebral injury is classified as mild or moderate (GCS score 10-15 points); Conservative treatment.
3. Within 72 hours after head injury, patients with stable and mentally handicapped mental state examination (MMSE) scores are lower than normal.
4. The legal representative and / or patient agree to participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

1. People who are known or suspected to be allergic to the test drug and its ingredients.
2. After the injury, drugs that improve cognitive function such as the prohibited drugs listed in the protocol have been used.
3. With a history of severe traumatic brain injury, a history of cerebrovascular accidents, and structural craniocerebral lesions.
4. With diseases such as speech and hearing impairment that cannot cooperate with the completion of cognitive function assessment.
5. A secondary brain injury occurred after the craniocerebral injury.
6. Those who need craniotomy or extraventricular drainage.
7. Combining with other serious large organ damage or serious complications may affect the test Life.
8. Patients with active epilepsy who had seizures within 1 year.
9. Patients with severe liver and kidney disease.
10. Complicated with severe heart disease, lung disease, blood and hematopoietic diseases, gastrointestinal disease, serious or progressive disease.
11. Past or present with a malignant tumor
12. Combining neurological and mental disorders that make it impossible or unwilling to cooperate.
13. Women who are pregnant, breastfeeding or have a recent birth plan.
14. Researchers do not consider it appropriate to participate in the clinical trial.
15. Those who have participated in other clinical trials and used test drugs 3 months before the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 591 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
The difference of Loewenstein Occupational Therapy Cognitive Assessment (LOCTA) scores between baseline and 3 months after administration of drugs. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Tianjin Medical University, Tianjing, Tianjing, China

REFERENCES:
- [Derived] Liu T, Wang J, Zhao Z, Jiang W, Zhang M, Yu Y, Liu Y, Liu M, Chen L, Zhang H, Hong Y, Li B, Yu R, Ji H, Mi L, Zhao B, Lv C, Liu C, Zhang J, Jiang R; LOCATE Trial Investigators. Efficacy and safety of L-oxiracetam on cognitive function in patients with traumatic brain injury: a multicentre, randomised, double-blind, phase 3 clinical trial. Signal Transduct Target Ther. 2025 Dec 12;10(1):401. doi: 10.1038/s41392-025-02492-5. PMID 41381424
- [Derived] Liu T, Liu M, Nie M, Zhao Z, Liu X, Qian Y, Yu Y, Sha Z, Wu C, Yuan J, Jiang W, Lv C, Mi L, Tian Y, Zhang J, Jiang R. Effect of l-oxiracetam and oxiracetam on memory and cognitive impairment in mild-to-moderate traumatic brain injury patients: Study protocol for a randomized controlled trial. Aging Med (Milton). 2024 Jun 14;7(3):341-349. doi: 10.1002/agm2.12335. eCollection 2024 Jun. PMID 38975302